CLINICAL TRIAL: NCT05386472
Title: A PHASE 1, OPEN-LABEL STUDY TO EVALUATE THE PHARMACOKINETICS, SAFETY, AND TOLERABILITY OF ORALLY ADMINISTERED NIRMATRELVIR/RITONAVIR IN PREGNANT WOMEN WITH MILD-TO-MODERATE COVID-19
Brief Title: A Study to Learn About the Study Medicine (Nirmatrelvir Plus Ritonavir) in Pregnant Women With COVID-19
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The trial prematurely terminated due to the inability to recruit the planned number of subjects. The decision to terminate the trial was not based on any safety concerns.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C4671035; NCT05386472 (Registry Identifier: ClinicalTrials.gov)
Record Dates: First submitted 2022-05-20; First posted 2022-05-23 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: COVID-19
Keywords: Severe acute respiratory syndrome coronavirus 2 (SARS-Cov-2); Pregnancy; Paxlovid; Nirmatrelvir
MeSH Terms: conditions — COVID-19 | interventions — nirmatrelvir; Ritonavir

STUDY DESIGN:
Masking Description: (Open Label)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort 1 (Experimental): Pregnant women in their second trimester
  Interventions: Drug: nirmatrelvir; Drug: ritonavir
- Cohort 2 (Experimental): Pregnant women in their third trimester
  Interventions: Drug: nirmatrelvir; Drug: ritonavir
- Cohort 3 (Experimental): Non-pregnant women
  Interventions: Drug: nirmatrelvir; Drug: ritonavir

INTERVENTIONS:
Drug: nirmatrelvir — Nirmatrelvir (tablets) administered by mouth every 12 hours for 5 days (10 doses total)
  Other Names: PF-07321332
Drug: ritonavir — Ritonavir (capsules) administered by mouth every 12 hours for 5 days (10 doses total)

SUMMARY:
The purpose of this clinical trial is to learn about how study medicine (Paxlovid, which contains nirmatrelvir and ritonavir) is changed and eliminated from the body, as well as its safety, and the extent to which side effects can be tolerated for treatment of pregnant women with mild or moderate COVID-19 compared to non-pregnant women with mild or moderate COVID-19.

This study is seeking participants who:

* are expecting a healthy baby and are in their second or third trimester pregnancy and have mild or moderate COVID-19
* are not pregnant and have mild or moderate COVID-19.

All participants in this study will take Paxlovid by mouth every 12 hours for 5 days. We will study the experiences of people receiving the study medicine. This will help us decide if the study medicine is safe.

All participants will take part in this study for at least 34 days; pregnant participants will take part until their delivery, so that the study duration may be up to 6 months, depending on their delivery date.

During this time, participants will have 7to 8 visits and, if pregnant, a visit at delivery. Around 2 to 3 visits and the delivery visit will be done in person (at the clinic or at the participant's home). The other 5 visits may be done over the phone, unless in-person visit is necessary as decided by the doctor. Blood samples will be collected on the first 4 to 5 study visits (and at other study visits, if necessary).

ELIGIBILITY:
Inclusion Criteria:

* All cohorts: Mild-to-moderate COVID-19 infection confirmed in sample collected ≤5 days prior to enrollment; onset within 5 days prior to enrollment and presence of ≥1 sign/symptom on the day of enrollment.
* Cohorts 1&2: Expecting single baby; Pregnant in 2nd trimester, 14 0/7 to 27 6/7 weeks of gestational age (Cohort 1) or 3rd trimester, ≥28 0/7 and ≤34 6/7 weeks of gestational age (Cohort 2), by ultrasound.
* All cohorts: Otherwise healthy participants who are determined by medical history, physical examination, and clinical judgment to be appropriate for inclusion in the study

Exclusion Criteria:

* All cohorts: Current need for hospitalization or anticipated need for hospitalization in the clinical opinion of the site investigator.
* Cohorts 1&2: Prior/current major condition or illness of mother/fetus substantially increasing risk of study participation/completion or impacting pregnancy/fetal outcomes in investigator's judgement.
* All cohorts: Current use of any medications that are highly dependent on CYP3A4 for clearance, and which are contraindicated in combination with nirmatrelvir/ritonavir.
* All cohorts: Has received or is expected to receive monoclonal antibody treatment, convalescent COVID-19 plasma, or anti-viral treatment (eg, molnupiravir) for the current SARSCoV-2 infection.
* All cohorts: Participants with moderate to severe kidney impairment

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Pregnant and non-pregnant females
Enrollment: 25 (Actual)
Dates: Start 2022-06-22 (Actual); Primary Completion 2025-03-26 (Actual); Study Completion 2025-05-12 (Actual)

PRIMARY OUTCOMES:
Apparent Oral Clearance (CL/F) | Day 1: 1-3 hour post-dose; Day 3: 4-8 hour post-dose; Day 4: 8 to less than 12 hour post dose; Day 5: 2-4 hour, 6-8 hour, 10 to less than 12 hour post dose.
Apparent Volume of Distribution (Vz/F) | Day 1: 1-3 hour post-dose; Day 3: 4-8 hour post-dose; Day 4: 8 to less than 12 hour post dose; Day 5: 2-4 hour, 6-8 hour, 10 to less than 12 hour post dose.
Area Under the Curve From Time Zero to End of Dosing Interval (AUCtau) | Day 1: 1-3 hour post-dose; Day 3: 4-8 hour post-dose; Day 4: 8 to less than 12 hour post dose; Day 5: 2-4 hour, 6-8 hour, 10 to less than 12 hour post dose.
Maximum Observed Plasma Concentration (Cmax) | Day 1: 1-3 hour post-dose; Day 3: 4-8 hour post-dose; Day 4: 8 to less than 12 hour post dose; Day 5: 2-4 hour, 6-8 hour, 10 to less than 12 hour post dose.
Plasma Decay Half-Life (t1/2) | Day 1: 1-3 hour post-dose; Day 3: 4-8 hour post-dose; Day 4: 8 to less than 12 hour post dose; Day 5: 2-4 hour, 6-8 hour, 10 to less than 12 hour post dose.
Observed Plasma Trough Concentration (Ctrough) | Day 1: 1-3 hour post-dose; Day 3: 4-8 hour post-dose; Day 4: 8 to less than 12 hour post dose; Day 5: 2-4 hour, 6-8 hour, 10 to less than 12 hour post dose.
Incidence of Treatment Emergent Adverse Events (TEAEs) | Baseline up through Day 34
Incidence of TEAEs, SAEs, and AEs leading to discontinuations | Baseline up through end of treatment (Day 5/Day 6)

SECONDARY OUTCOMES:
Number of participants with delivery at medical facility | At delivery of the baby
Number of participants with delivery at home | At delivery of the baby
Number of participants with delivery at other location | At delivery of the baby
Number of participants with caesarean section delivery | At delivery of the baby
Number of participants with vaginal delivery | At delivery of the baby
Number of participants with complications during delivery | At delivery of the baby
Number of full-term live deliveries | At delivery of the baby
Number of premature live deliveries | At delivery of the baby
Number of participants with stillbirths | At delivery of the baby
Number of participants with spontaneous abortions | At delivery of the baby
Number of participants with induced/elective abortions | At delivery of the baby
Number of participants with unknown delivery | At delivery of the baby
Number of aborted or stillborn fetuses with abnormal findings upon gross visual inspection | At delivery of the baby
Gestational age of newborn infants | At birth
Number of neonates with congenital malformation/anomaly or other neonatal problem | At birth
Body weight of newborn infants | At birth
Body length of newborn infants | At birth
Head circumference of newborn infants | At birth
Incidence of SAEs in newborn infants | Birth through 24 hours after birth or until Study Day 34 (whichever is later)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (12):
- United States (12):
  - University of Alabama at Birmingham/Center for Women's Reproductive Health, Birmingham, Alabama
  - Beautiful Minds Clinical Research Center, Cutler Bay, Florida
  - Omega Research Debary, DeBary, Florida
  - Omega Research Orlando, Orlando, Florida
  - Santos Research Center, Tampa, Florida
  - Clinical Research Prime, Idaho Falls, Idaho
  - Boeson Research MSO, Missoula, Montana
  - Origin Health, Missoula, Montana
  - Maximos Ob/Gyn, League City, Texas
  - University of Utah, Salt Lake City, Utah
  - University of Utah Clinical Neuroscience Center, Salt Lake City, Utah
  - University of Utah Hospital, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C4671035